CLINICAL TRIAL: NCT03852602
Title: Preemptive Analgesia for Postoperative Pain Control for Dental Treatment Under General Anesthesia in Children
Brief Title: Preemptive Analgesia for Postoperative Pain Control for Dental Treatment Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Collaborators: Inonu University (Other)
Responsible Party: Principal Investigator, Sultan KELES, Assist. Prof.Dr., Aydin Adnan Menderes University
Other Study IDs: 2019-18
Record Dates: First submitted 2019-02-18; First posted 2019-02-25 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Control: Analgesic application15 minutes before the end of the treatment will constitute the control group.
  Interventions: Drug: Control
- Group preemptive: Patients who underwent analgesic 15 minutes after the induction of general anesthesia .
  Interventions: Drug: Preemptive Analgesics

INTERVENTIONS:
Drug: Preemptive Analgesics — Analgesic application15 minutes before the treatment
  Groups: Group preemptive
Drug: Control — Analgesic application15 minutes before the end of the treatment
  Other Names: Preventive analgesic
  Groups: Group Control

SUMMARY:
The aim of this study was to compare the analgesic-treated children with analgesic prior to the treatment and to compare the postoperative analgesic needs of children undergoing dental treatment under general anesthesia.

DETAILED DESCRIPTION:
The investigator's study included patients who were admitted to Inonu University and Adnan Menderes University, Faculty of Dentistry, Department of Pediatric Dentistry in 2019 and decided to perform dental treatment under general anesthesia. Patients 1 to 7 years of age with dental treatment between February 28 and June 1, 2019 will be included.

Patients who underwent analgesic 15 minutes after the induction of general anesthesia from the patients, and those who made painkillers 15 minutes before the end of the treatment will constitute the control group. Paracetamol 15 mg / kg IV will be given in 50 ml of saline.

The demographic data of the children to be included in the study such as age, gender, type of dental intervention, duration of operation, postoperative pain scores, recovery times will be recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* To be treated under general anesthesia
* No systemic disease
* To have at least one painful dental procedure in the upper and lower jaw (pulpectomy, pulpotomy

Exclusion Criteria:

* Patients with mental or physical disabilities of any disease
* Patients who have not undergone painful dental intervention under general anesthesia

Ages: 3 Years to 7 Years | Sex: All
Age Groups: Child
Study Population: Children who will be treated under general anesthesia because of lack of chairside cooperation.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Postoperative dental pain | An average of 24 hours postoperatively
  Wong-Baker faces Scale is validated for children aged 3 to 7 years, includes six cartoon faces corresponding to scores 0-5 (0=no hurt, 1= hurts a little bit, 2= hurts a little more, 3=hurts even more, 4= hurts a whole lot, 5=hurts worst).

CONTACTS AND LOCATIONS:
Overall Officials: Sultan Keles, Dr., Study Chair — Aydin Adnan Menderes University
Locations (1):
- Sultan KELES, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Study will be conducted and then will be published.

REFERENCES:
- [Background] Kharouba J, Hawash N, Peretz B, Blumer S, Srour Y, Nassar M, Sabbah M, Safadi A, Khorev A, Somri M. Effect of intravenous paracetamol as pre-emptive compared to preventive analgesia in a pediatric dental setting: a prospective randomized study. Int J Paediatr Dent. 2018 Jan;28(1):83-91. doi: 10.1111/ipd.12311. Epub 2017 Jun 15. PMID 28618198